CLINICAL TRIAL: NCT02103998
Title: Phase III Study of Thyroid Hormones in Prematures
Brief Title: Study of Thyroid Hormones in Prematures
Acronym: THOP2
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: not funded by NIH
Sponsor: New York Medical College (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Edmund F LaGamma, MD, Professor of Pediatrics, New York Medical College
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: THOP2 - NYMC - CCC
Record Dates: First submitted 2013-05-02; First posted 2014-04-04 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Transient Hypothyroxinemia of Prematurity (THOP)
Keywords: extremely low gestational age neonate; hypothyroxinemia of prematurity; brain development; cerebral palsy; cognitive dealy
MeSH Terms: conditions — Cerebral Palsy | interventions — Potassium Iodide; WW Domain-Containing Oxidoreductase; Thyroxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- T4 + KI (Experimental): Continuous infusion of 4 µg/Kg/day T4 with 30 µg/Kg/day oral potassium iodide (KI) for 42 days
  Interventions: Drug: thryoid hormone T4 + oral potassium iodide (KI) for 42 days
- D5W - 5% dextrose water (Placebo Comparator): Receive the same volume as study drug but as D5W placebo
  Interventions: Drug: D5W - 5% dextrose water

INTERVENTIONS:
Drug: thryoid hormone T4 + oral potassium iodide (KI) for 42 days — Continuous infusion of 4 µg/Kg/day T4 with 30 µg/Kg/day oral potassium iodide (KI) for 42 days
  Other Names: levothyroxin; postassium iodide
  Arms: T4 + KI
Drug: D5W - 5% dextrose water — Equivalent volume of infusion as study drug
  Other Names: Standard hospital pharmacy solution
  Arms: D5W - 5% dextrose water

SUMMARY:
The investigators hypothesize that continuous infusion of 4 µg/Kg/day T4 with 30 µg/Kg/day oral potassium iodide (KI) for 42 days from birth will reduce by 30% or more (from an estimated 30% to 21%) the proportion of extremely low gestational age subjects with a composite endpoint of "cerebral palsy (CP) or a Bayley III Composite Cognitive Score < 85" at 36 months corrected postnatal age (CA).

DETAILED DESCRIPTION:
This study is a Phase III multicenter, masked, placebo controlled randomized clinical trial (RCT) of thyroid hormone supplementation in premature infants. Survival for extremely low gestational age neonates (ELGAN; 24 - 28 weeks) has risen to >80% over the past 40 years yet cognitive delays or cerebral palsy (CP) still affect 30% of survivors. Since more than 25,000 ELGANs are born each year in the United States, a major priority in newborn medicine must be to translate the gains in survival into gains in healthy survival without the current high frequency of impairments. Transient hypothyroxinemia of prematurity (THOP) occurs in 50% of ELGANs and is strongly associated as an independent risk factor with lower IQ scores, behavioral abnormalities and CP in ELGANs. Prior evidence suggested a benefit from replacement therapy but studies were underpowered to prove this. The current project extends the findings of our Phase 1 trial (THOP1; R01-NS45109) where four thyroid hormone regimens were tested. We showed that continuous infusion of 4 µg/Kg/day thyroxine x 42d could safely correct transient hypothyroxinemia without markedly lowering TSH - creating a "biochemical euthyroid" state. THOP2 is designed to test the primary hypothesis that compared to placebo, thyroid hormone supplementation from birth will reduce from 30% to 21% the proportion of subjects with a composite endpoint of "CP or a Bayley III Cognitive Score < 85." A Secondary hypothesis is that hormone treatment will improve other measures of cognitive and executive function or attention as assessed by: i) Bayley III Parent Interview for Adaptive Behavior and the BRIEF-P (Behavioral Rating Inventory of Executive Function-Preschool Version) and ii) the frequency of screening positive on the Modified Checklist for Autism in Toddlers (M-CHAT). We plan to enroll 1,224 subjects over a 19.8 month period at 14 centers to obtain 388 surviving toddlers at 36 months corrected age in each of two arms. The current application describes the scientific basis of the proposed overall clinical trial; it is linked to a cluster application creating a Data Monitoring and Analysis Coordinating Center (DCC) at Michigan State University (MSU). The additional societal cost from CP in an affected person's lifetime is estimated at $1 million; the costs of mental retardation are even higher. If this trial shows that an inexpensive intervention can reduce the risks of CP and mental retardation by 30% in ELGANs, we estimate the overall savings from preventing more than 2,000 such cases (9% of 25,000) at about $2 billion per year.

ELIGIBILITY:
Inclusion Criteria:

1. Neonates 24 0/7 to 27 6/7 weeks gestational age
2. inborn or transferred; < 24 hours old

Exclusion Criteria:

1. Maternal or congenital thyroid disease or
2. Maternal substance abuse by history at the time of birth (heroin or cocaine)
3. Major congenital or surgical malformations of neonate
4. Known chromosomal anomalies detected by antepartum testing or direct physical examination
5. Absence of parental consent or treating physician assent
6. A concurrent clinical trial with another randomized drug
7. Death expected < 48h vi) Another concern by the treating physician that either mandates or prohibits study treatment such as known adverse drug interaction
8. mother < 18 years old at delivery

Ages: 1 Hour to 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Compare incidence of a COMPOSITE endpoint of "cerebral palsy (CP) or a Bayley III Composite Cognitive Score < 85" at 36 months corrected postnatal age (CA). | 36 months
  Bayley III Cognitive Score and a standardize ELGAN-type neurological exam (Kuban) plus a Palisano assessment of function

SECONDARY OUTCOMES:
Compare measures of cognitive and executive function and attention. | 36 months corrected age
  As assessed by the following tests:
  1. The mean scores of the Bayley III Parent Interview for Adaptive Behavior and the BRIEF-P (Behavioral Rating Inventory of Executive Function-Preschool Version).
  2. The frequency of screening positive on the Modified Checklist for Autism in Toddlers (M-CHAT).

CONTACTS AND LOCATIONS:
Overall Officials: Edmund F La Gamma, MD, Principal Investigator — New York Medical College
Locations (1):
- Maria Fareri Childrens Hospital, Valhalla, New York, United States

REFERENCES:
- [Result] La Gamma EF, van Wassenaer AG, Ares S, Golombek SG, Kok JH, Quero J, Hong T, Rahbar MH, de Escobar GM, Fisher DA, Paneth N. Phase 1 trial of 4 thyroid hormone regimens for transient hypothyroxinemia in neonates of <28 weeks' gestation. Pediatrics. 2009 Aug;124(2):e258-68. doi: 10.1542/peds.2008-2837. Epub 2009 Jul 5. PMID 19581264